CLINICAL TRIAL: NCT07104799
Title: A Phase I Study to Evaluate the Safety and Maximum Tolerated Dose of Momelotinib Durind and Following Hematopoietic Cell Transplantation for Patients With Myelofibrosis
Brief Title: Momelotinib During and After HCT in Myelofibrosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Gabriela Hobbs, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-501
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Myelofibrosis; Hematopoietic Cell Transplantation (HCT)
Keywords: myelofibrosis; allogeneic hematopoietic cell transplantation (HCT); HCT
MeSH Terms: conditions — Primary Myelofibrosis | interventions — N-(cyanomethyl)-4-(2-((4-(4-morpholinyl)phenyl)amino)-4-pyrimidinyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Momelotinib + Standard of Care (SOC) Hematopoietic Cell Transplantation (HCT) (Experimental): Momelotinib will be administered orally once daily at a pre-determined dose starting 7 days before standard of care (SOC) hematopoietic cell transplantation (HCT) and for up to 1 year after HCT, for a total of 13 28-day cycles. Participants will receive SOC HCT and HCT treatment including: reduced intensity conditioning (RIC) regimen before HCT (Fludarabine, Mephalan), and tacrolimus and methotrexate after HCT, all administered according to SOC.
  Interventions: Drug: Momelotinib

INTERVENTIONS:
Drug: Momelotinib — Administered orally once per day during each 28-day cycle. This will start on day -7 (7 days before HCT) and continue for up to 13 cycles. Dose cohorts (100 mg daily, 150 mg daily, 200 mg daily) will be investigated in the peri-transplant period. Once participants have achieved hematopoietic recovery and are at least Day 21 after HCT, participants will increase the dose to 200 mg daily.
  Other Names: GSK3070785

SUMMARY:
This is a single-center, open-label, phase I study to determine the safety and tolerability of momelotinib in patients with myelofibrosis during and after hematopoietic cell transplantation (HCT).

DETAILED DESCRIPTION:
The purpose of this study is to test the safety, effects, and recommended dose of an investigational drug, momelotinib, during and after undergoing allogeneic HCT. This study will enroll up to 28 participants with myelofibrosis that are planned to undergo standard of care allogeneic hematopoietic cell transplantation (HCT). Participants may receive momelotinib or other JAK inhibitors prior to HCT and may adjust momelotinib dosing per protocol as follows: Multiple dose cohorts (100 mg daily, 150 mg daily and 200 mg daily) will be investigated in the peri-transplant period. Participants not previously on momelotinib will begin this drug at the initiation of conditioning therapy (Day -7 from HCT). Once participants have achieved hematopoietic recovery and are at least Day 21(cycle 2 day 1) after HCT, participants, receiving lower doses will increase the dose to 200 mg daily. Patients will remain on momelotinib for a total of 13 cycles (28 days per cycle, until approximately 1 year after transplant). After HCT, participants will be followed for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have pathologically confirmed primary myelofibrosis (PMF) according to WHO criteria or secondary myelofibrosis as defined by the IWG-MRT criteria.

  * Intermediate-2/ high-risk disease as per Dynamic IPSS (DIPSS) Plus criteria OR
  * Intermediate-1 risk disease with at least one of the following unfavorable features known to impact the survival adversely

    * Red cell transfusion dependency
    * Unfavorable Karyotype
    * Platelet count ≤100 x 10^9/L
    * Presence of a high risk molecular marker associated with worsened overall survival (ASXL1, EZH2, IDH1/2, SRSF2, U2AF1, p53)
* Participants do not have to be receiving treatment with JAK inhibitors for MF at the time of enrollment. If participants are receiving JAK inhibitor therapy with agents other momelotinib, participants must agree to be switched to momelotinib to begin Cycle 1 Day 1 on Day -7 from HCT (at the initiation of conditioning).
* Age >18 years
* Participants must be designated to undergo allogeneic HCT with:

  * reduced intensity conditioning regimen, and
  * peripheral blood stem cells as a graft source
* Participants who will undergo HCT from the following donor types are eligible:

  * 6/6 (HLA-A, B, DR) fully matched related donor or
  * 8/8 (HLA-A, B, DR, C) fully matched unrelated donor. Matching in the unrelated setting must be at the allele level
* ECOG performance status ≤2 (Karnofsky ≥60%)
* The effects of momelotinib on the developing human fetus are unknown. Female patients of childbearing potential must have a negative pregnancy test, as measured by serum or urine testing. Women of childbearing potential: must agree to use highly effective contraception prior to the initial dose/start of the first treatment, during the study, and for at least 1 week after the last dose of momelotinib.

Male participants with women of child bearing potential partners must agree to use one of the forms of medically acceptable birth control at start of the first treatment, during the study, and for at least 6 months after the last dose. See Exclusion Criteria for effective contraception and birth control.

- Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Known intolerance or hypersensitivity to any JAK inhibitor, including ruxolitinib, fedratinib, pacritinib, momelotinib or any other JAK inhibitor, its metabolites or formulation excipients.
* Has had any major surgery within 28 days prior to randomization
* Has received treatment with an investigational agent within 4 weeks of the first dose of study intervention
* Has received immunosuppressive agents within 28 days
* Prior allogeneic transplant for any hematopoietic disorder
* Had accelerated phase or leukemic transformation (≥10% blasts in bone marrow any time prior to HCT)
* Has an active, uncontrolled infection
* Has cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal/gastric varices, or persistent jaundice.
* Known diagnosis of active hepatitis B or hepatitis C.
* History of another malignancy(ies), unless:

  * the participant has been disease-free for at least 2 years and is deemed by the investigator to be at low risk of recurrence of that malignancy, or
  * the cancer has been deemed indolent with no progression over the last 2 years, and deemed by the investigator to be at low risk for further progression during the course of study and follow-up
  * the only prior malignancy was cervical cancer in situ and/or basal cell or squamous cell carcinoma of the skin
* Participants without normal organ function defined as follows:

  * AST (SGOT), ALT (SGPT) and Alkaline Phosphatase >3 × institutional Upper Limit of Normal (ULN)
  * Total bilirubin >1.5 mg/dL, with the exception of participants with Gilbert's Syndrome provided direct bilirubin is ≤1.5x ULN and participant otherwise meets entry criteria.
  * Calculated creatinine clearance ≤60 mL/min (Cockcroft-Gault formula)
  * Have current or a history of congestive heart failure New York Heart Association (NYHA) class 3 or 4, or any history of documented diastolic or systolic dysfunction (LVEF < 40%, as measured by MUGA scan or echocardiogram) or clinically significant arrhythmia not controlled by standard of care therapy.
* Not able to take oral medication or having any clinically significant gastrointestinal abnormalities that may alter absorption, e.g., malabsorption syndrome or major resection of the stomach and/or bowels.
* Grade 2 or greater peripheral neuropathy
* Pregnant or lactating women, or women planning to become pregnant or initiating breastfeeding.
* To exclude women of childbearing potential: who are unwilling or unable to practice highly effective contraception prior to the initial dose/start of the first treatment, during the study, and for at least 1 week after the last dose. Highly effective contraceptive measures include:

  * stable use of combined (estrogen and progestogen containing) hormonal contraception (oral, intravaginal, transdermal) or progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation initiated 2 or more menstrual cycles prior to screening;
  * intrauterine device (IUD); intrauterine hormone-releasing system (IUS);
  * sexual abstinence;
  * intercourse with vasectomized partner (provided that the male vasectomized partner is the sole sexual partner of the WOCBP study participant and that the vasectomized partner has obtained medical assessment of surgical success for the procedure).
* To exclude sexually active male participants with WOCBP partners who are unwilling to use the one of the following forms of medically acceptable birth control at start of the first treatment, during the study, and for at least 6 months after the last dose:

  * vasectomy with medical assessment of surgical success OR consistent use of a condom.
  * male participants must also agree not to donate sperm while receiving study drug and for at least 6 months after the last dose.
* Patients receiving strong CYP 3A4 inducers during study period
* Patients with major ABO mismatch donors only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Momelotinib | From start of study treatment (Day -7) through 28 days.
  MTD is defined as the highest dose level at which 0 or 1 of 6 patients experience a Dose Limiting Toxicity (DLT). Toxicities will be graded and documented according to NCI CTCAE version 5.0.

SECONDARY OUTCOMES:
Incidence of momelotinib-related toxicities | Day -7 through 30 days after end of treatment (up to 394 days)
  Toxicity will be categorized and graded per NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0 criteria.
Median Duration of Momelotinib Therapy | Day -7 through end of treatment, up to 364 days.
  Median duration of momelotinib therapy during and after allogeneic HCT will be calculated and is the duration of study treatment which divides the shortest 50% and longest 50% of treatment durations.
Median time to neutrophil engraftment | Day 0 (Day of HCT) through Day 60.
  Neutrophil engraftment will be defined as first of 3 successive days with an absolute neutrophil count of greater than or equal to 0.5 x 10^9/l after post-HCT nadir. Median time to neutrophil engraftment for participants receiving momelotinib during allogeneic HCT will be calculated.
Median time to platelet engraftment | Day 0 (Day of HCT) through Day 60.
  Platelet engraftment will be defined as first of 3 successive days with platelet count of greater than or equal to 20 x 10^9/l in the absence of platelet transfusion for 7 consecutive days. Median time to platelet engraftment for participants receiving momelotinib during allogeneic HCT will be calculated.
Time to red blood cell transfusion independence | Day 0 through end of treatment, up to 1 year.
  Transfusion independence is defined as clinical hematologic recovery requiring no transfusion in the past 7 days. The time from Day 0 to transfusion independence will be reported.
Cumulative incidence of primary graft failure | Day 0 through Day 60.
  Primary graft failure will be defined as lack of achievement of an absolute neutrophil count of greater than or equal to 0.5 x 10^9/l by Day +30 after HCT with associated pancytopenia. Incidence of primary graft failure in participants receiving momelotinib during and after allogeneic HCT will be reported.
Cumulative incidence of acute graft-versus-host disease (GVHD) | Day 0 through 2 years after HCT
  Clinical stage and grade of acute graft-versus-host-disease (GVHD) is based on MAGIC Criteria. The incidence of acute GVHD grade II-IV and grade III-IV will be estimated for each treatment group using the cumulative incidence estimate, treating death prior to acute GVHD as a competing event. Incidence of acute GVHD in participants receiving momelotinib during and after allogeneic HCT will be reported.
Cumulative incidence of chronic graft-versus-host disease (GVHD) | Day 0 through 2 years after HCT
  Chronic GVHD will be assessed as per the 2014 National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease. The incidence of chronic GVHD will be estimated for each treatment group using the cumulative incidence estimate, treating death prior to chronic GVHD as a competing event.
Incidence of Non-relapse mortality (NRM) | Day -7 through 2 years post HCT.
  Clinical response is evaluated using the using the Revised IWG-MRT, ELN response criteria for Myelofibrosis, and recently defined endpoints for MF based on recently defined consensus criteria. The incidence of non-relapse mortality (NRM) will be estimated for each treatment group using the cumulative incidence estimate, treating disease relapse or progression as a competing event. NRM will be estimated in the context of a competing risks framework. Gray test will be used for group comparison of cumulative incidence of NRM.
Progression-free survival (PFS) | Day -7 through 2 years post HCT.
  Clinical response is evaluated using the using the Revised IWG-MRT, ELN response criteria for Myelofibrosis, and recently defined endpoints for MF based on recently defined consensus criteria. Progression-free survival is defined as the time from first dose of study drug to the earlier of disease relapse or death due to any cause. Participants alive and progression-free are censored at the date of last disease evaluation.
Overall survival (OS) | Day -7 through 2 years post HCT.
  Overall Survival is defined as the time from first dose of study drug to the date of death due to any cause. Participants who are alive at the analysis / cutoff date will be censored at the last contact date. OS will be estimated using the Kaplan-Meier method and compared using log-rank test.
GVHD-free, relapse-free survival (GRFS) | Day -7 through 2 years post HCT
  GVHD, relapse-free survival is defined as the time from first dose of study drug to the earlier of grade III-IV acute GVHD, chronic GVHD requiring systemic immune suppression, leukemia relapse or death due to any cause. Participants alive and without one of these three events are censored at the date of last disease evaluation. GRFS will be estimated using the Kaplan-Meier method and compared using log-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Hobbs, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: Gabriela Hobbs, MD, ghobbs@mgb.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation